CLINICAL TRIAL: NCT07342413
Title: A Single-center Prospective Double-Blind, Split-Body, Randomized Clinical Study Comparing Glycerin With 1% Lidocaine and Epinephrine Versus Glycerin With 1% Lidocaine Without Epinephrine for the Sclerotherapy of Leg Telangiectasias
Brief Title: Study Comparing Glycerin With 1% Lidocaine and Epinephrine Versus Glycerin With 1% Lidocaine Without Epinephrine for the Sclerotherapy of Leg Telangiectasias
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Sclero-Epi-2025
Record Dates: First submitted 2026-01-13; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Leg Veins
MeSH Terms: interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A Right Leg Treated with glycerin compounded 1% lidocaine and epinephrine (Active Comparator): Subjects will be treated with foamed sodium tetradecyl sulfate (STS) to both legs. Four weeks later subjects left leg will be treated with glycerin compounded with 1% lidocaine, and right leg will be treated with glycerin compounded with 1% lidocaine and epinephrine.
  Interventions: Drug: Right leg treated with Glycerin compounded with 1% Lidocaine and Epinephrine
- Group B Left Leg Treated with glycerin compounded 1% lidocaine and epinephrine (Sham Comparator): Subjects will be treated with foamed sodium tetradecyl sulfate (STS) to both legs. Four weeks later subjects right leg will be treated with glycerin compounded with 1% lidocaine, and left leg will be treated with glycerin compounded with 1% lidocaine and epinephrine.
  Interventions: Drug: Left leg treated with Glycerin compounded with 1% Lidocaine and Epinephrine

INTERVENTIONS:
Drug: Right leg treated with Glycerin compounded with 1% Lidocaine and Epinephrine — Right leg treated with glycerin compounded with 1% lidocaine and epinephrine
  Arms: Group A Right Leg Treated with glycerin compounded 1% lidocaine and epinephrine
Drug: Left leg treated with Glycerin compounded with 1% Lidocaine and Epinephrine — Left leg treated with glycerin compounded with 1% lidocaine and epinephrine
  Arms: Group B Left Leg Treated with glycerin compounded 1% lidocaine and epinephrine

SUMMARY:
The primary objective is to compare physician-assessed clearance of telangiectatic veins between treatment legs using the Physician Global Aesthetic Improvement Scale (PGAIS). Secondary objectives include assessment of procedural pain, safety outcomes, and patient satisfaction.

DETAILED DESCRIPTION:
This is a prospective, double-blind, split-body, randomized, controlled pilot study enrolling twenty (20) adult subjects.

Subjects with reticular veins (≥1 mm) will first undergo pre-treatment with foamed sodium tetradecyl sulfate (STS) using the investigator's standard technique. Subjects without reticular veins will proceed directly to telangiectasia treatment. At a subsequent treatment visit approximately four weeks later, subjects will undergo split-leg sclerotherapy for telangiectatic veins (<1 mm), with one leg randomized to receive glycerin compounded with 1% lidocaine, and the contralateral leg randomized to receive glycerin compounded with 1% lidocaine and epinephrine (1:100,000).

Each subject will serve as their own control.Both the treating investigator and the subject will remain blinded to treatment allocation. Efficacy assessments will be performed by a non-treating, blinded investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 20-75years.
2. Fitzpatrick skin types I-VI.
3. Presence of lower extremity telangiectatic veins (<1 mm) suitable for sclerotherapy (reticular veins ≥1 mm can be present but are not required).
4. Duplex ultrasonography negative for saphenous vein reflux in both legs.
5. Willing to undergo split-leg randomization (CG + 1% lidocaine vs CG + 1% lidocaine with epinephrine 1:100,000).
6. Willing and able to comply with all study procedures, including standardized photography, in-person evaluations by a non-treating physician investigator, Day 90 follow-up assessments, and post-treatment compression therapy consisting of graduated 30-40 mmHg stockings worn 24 hours/day for 1 week following treatment.
7. Subject with no known history of coagulopathy/platelet disorders (eg., hemophilia, von Willebrand disease) or liver disease/cirrhosis
8. Subject with no history of hypercoagulable disorder such as pulmonary embolism, deep vein thrombosis, factor V Leiden mutation, Protein C or S deficiency, antiphospholipid syndrome, or active malignancy
9. Subjects in good general health as determined by the investigator's judgment and medical history.
10. Participants must be willing to provide written informed consent and sign a photography release for research and potential publication. Subjects must also agree to complete all study visits and procedures.
11. Willing to avoid new lower-extremity aesthetic/vascular treatments (e.g., sclerotherapy, vascular lasers) and agree to avoid self-tanners or spray tans on the legs during the study period.
12. Negative urine pregnancy test result at the time of study entry and all subsequent visits (if applicable)
13. Subjects of childbearing potential must agree to use an effective method of birth control during the entire course of the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment.

    1. Acceptable forms of birth control are: oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine device/coil, bilateral tubal ligation, double-barrier methods (e.g., sponge, spermicide, or condoms). Abstinence and/or vasectomized partner must agree to a second acceptable method of birth control (double-barrier) should the subject become sexually active.
    2. A female is considered of non-childbearing potential if she is: postmenopausal (no menses for at least 12 months/≥ 12 months of amenorrhea without another medical cause), without a uterus (hysterectomy) and/or both ovaries (oophorectomy).

Exclusion Criteria:

1. Positive duplex ultrasonography demonstrating saphenous vein reflux.
2. Prior sclerotherapy or vascular laser treatment to the lower extremities within the past 6 months prior to screening/baseline
3. History of ulceration, thrombophlebitis, or deep vein thrombosis (DVT) in the lower extremities.
4. Active infection, open wounds, or inflammatory dermatoses (e.g., eczema, psoriasis, dermatitis) in the treatment area.
5. Known allergy or hypersensitivity to lidocaine, epinephrine, or glycerin.
6. Any uncontrolled systemic condition that may increase risk or interfere with study participation (e.g., poorly managed diabetes, thyroid dysfunction, cardiovascular disease).
7. Pregnancy, intent to become pregnant during the study period, or current breastfeeding.
8. Clinically significant psychiatric or psychological conditions that, in the opinion of the investigator, may interfere with compliance or interpretation of results
9. Participation in another clinical study within 30 days prior to enrollment of this study or during this study.
10. Unwillingness to refrain from additional lower extremity aesthetic/vascular treatments (e.g., sclerotherapy, vascular lasers, self-tanning) from the screening/baseline visit through the end of study.
11. Unwillingness to follow a wash-out period of 4 weeks prior to screening for self-tanner application.
12. Unwillingness to refrain from self-tanner application for 1 month prior to any visits.
13. Unwillingness or inability to comply with post-treatment compression therapy consisting of graduated 30-40 mmHg stockings worn 24 hours/day for 1 week following treatment

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Physician Global Aesthetic Improvement Scale PGAIS | Day 90
  Please rate right leg veins:
  Circle One
  * 2 Much Improved
  * 1 Improved 0 No Change
    * 1 Worse
    * 2 Much Worse
  Please rate left leg veins:
  Circle One
  * 2 Much Improved
  * 1 Improved 0 No Change
    * 1 Worse
    * 2 Much Worse

SECONDARY OUTCOMES:
Patient Satisfaction Likert Score for vein improvement | Day 90
  Please rate right leg veins:
  Circle One
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
  Please rate left leg veins:
  Circle One
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
Visual Analog Pain Scale Post Treatment | Day 1 and Day 30
  Please rate pain for right leg:
  Circle One 0 No Pain 1-3 Mild 4-6 Moderate to Severe 7-9 Very Severe 10 Worst Pain Possible
  Please rate pain for left leg:
  Circle One 0 No Pain 1-3 Mild 4-6 Moderate to Severe 7-9 Very Severe 10 Worst Pain Possible

CONTACTS AND LOCATIONS:
Locations (1):
- West Dermatology Research Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided